CLINICAL TRIAL: NCT04453202
Title: A Randomized, Double-blind, Placebo-controlled Phase 2a Study to Evaluate a Range of Dose Levels of an Ad26.RSV.preF-based Vaccine in Adults Aged 60 Years and Older
Brief Title: A Study to Evaluate a Range of Dose Levels of an Adenovirus Serotype 26 (Ad26.RSV.preF)-Based Vaccine in Older Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CR108835; VAC18193RSV2005 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2020-06-29; First posted 2020-07-01 (Actual); Results first posted 2023-10-03 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Healthy
MeSH Terms: interventions — Respiratory Syncytial Virus Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Cohort 1 Group 1: RSV Vaccine (Experimental): Participants will receive a single intramuscular (IM) injection of an Ad26-based RSV vaccine on Day 1.
  Interventions: Biological: RSV Vaccine
- Cohort 1 Group 2: RSV Vaccine (Experimental): Participants will receive a single IM injection of an Ad26-based RSV vaccine (low dose 1) on Day 1.
  Interventions: Biological: RSV Vaccine
- Cohort 1 Group 3: RSV Vaccine (Experimental): Participants will receive a single IM injection of an Ad26-based RSV vaccine (low dose 2) on Day 1.
  Interventions: Biological: RSV Vaccine
- Cohort 1 Group 4: RSV Vaccine (Experimental): Participants will receive a single IM injection of an Ad26-based RSV vaccine (low dose 3) on Day 1.
  Interventions: Biological: RSV Vaccine
- Cohort 1 Group 5: Placebo (Placebo Comparator): Participants will receive IM injection of placebo on Day 1.
  Interventions: Other: Placebo
- Cohort 2 Group 6: RSV Vaccine (Experimental): Participants will receive a single IM injection of an Ad26-based RSV vaccine on Day 1.
  Interventions: Biological: RSV Vaccine
- Cohort 2 Group 7: RSV Vaccine (Experimental): Participants will receive a single IM injection of an Ad26-based RSV vaccine (high dose 1) on Day 1.
  Interventions: Biological: RSV Vaccine
- Cohort 2 Group 8: Placebo (Placebo Comparator): Participants will receive IM injection of placebo on Day 1.
  Interventions: Other: Placebo
- Cohort 3 Group 9: RSV Vaccine (Experimental): Participants will receive a single IM injection of an Ad26-based RSV vaccine on Day 1.
  Interventions: Biological: RSV Vaccine
- Cohort 3 Group 10: RSV Vaccine (Experimental): Participants will receive a single IM injection of an Ad26-based RSV vaccine (high dose 2) on Day 1.
  Interventions: Biological: RSV Vaccine
- Cohort 3 Group 11: Placebo (Experimental): Participants will receive IM injection of placebo on Day 1.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: RSV Vaccine — Participants will receive a single IM injection of an Ad26-based RSV vaccine on Day 1.
  Arms: Cohort 1 Group 1: RSV Vaccine; Cohort 1 Group 2: RSV Vaccine; Cohort 1 Group 3: RSV Vaccine; Cohort 1 Group 4: RSV Vaccine; Cohort 2 Group 6: RSV Vaccine; Cohort 2 Group 7: RSV Vaccine; Cohort 3 Group 10: RSV Vaccine; Cohort 3 Group 9: RSV Vaccine
Other: Placebo — Participants will receive a single IM injection of placebo on Day 1.
  Arms: Cohort 1 Group 5: Placebo; Cohort 2 Group 8: Placebo; Cohort 3 Group 11: Placebo

SUMMARY:
The purpose of this study is to explore the dose-response relationship of immune responses induced by different dose levels of an Ad26.RSV.preF based vaccine (Cohort 1) and to assess the safety and reactogenicity of different dose levels of the Ad26.RSV.preF-based vaccine (Cohorts 2 and 3).

ELIGIBILITY:
Inclusion Criteria:

* In the investigator's clinical judgment, participants must be either in good or stable health. Participants may have underlying illnesses such as hypertension, type 2 diabetes mellitus, hyperlipoproteinemia, or hypothyroidism, as long as their signs and symptoms are stable and medically controlled in the judgment of the investigator. Participants will be included on the basis of medical history and of physical examination and vital signs performed at screening (all cohorts), and of physical examination and/or vital signs performed prevaccination on Day 1 (Cohorts 2 and 3)
* A woman must be postmenopausal (defined as no menses for 12 months without an alternative medical cause) and not intending to conceive by any methods
* Agree to not donate blood from the time of vaccination until 3 months after vaccination
* Have a body mass index (BMI) less than (<) 40 kilogram per meter square (kg/m^2)
* Be willing to provide verifiable identification and have means to be contacted and to contact the investigator during the study

Exclusion Criteria:

* Has a contraindication to intramuscular injection (IM) injections and blood draws (example, bleeding disorders)
* Known allergy or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine components (including any of the constituents of the study vaccine)
* History of chronic urticaria (recurrent hives), eczema, or atopic dermatitis
* Has hepatitis B or C infection, including history of treated hepatitis C infection
* Received an active RSV vaccine in a previous RSV vaccine study or an Ad26-vectored vaccine at any time prior to randomization

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2021-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (9):
- United States (9):
  - Optimal Research, San Diego, California
  - Clinical Research of South Florida, an AMR Company, Coral Gables, Florida
  - Heartland Research Associates, an AMR Company, El Dorado, Kansas
  - Optimal Research, Rockville, Maryland
  - The Center for Pharmaceutical Research (CPR), Kansas City, Missouri
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - Meridian Clinical Research - Omaha, Omaha, Nebraska
  - Tekton Research Inc., Yukon, Oklahoma
  - AMR New Orleans, Formerly New Orleans Center for Clinical Research - New Orleans, an AMR company, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] van Heesbeen R, Bastian AR, Omoruyi E, Rosen J, Comeaux CA, Callendret B, Heijnen E. Immunogenicity and safety of different dose levels of Ad26.RSV.preF/RSV preF protein vaccine in adults aged 60 years and older: A randomized, double-blind, placebo-controlled, phase 2a study. Vaccine. 2024 Dec 2;42(26):126273. doi: 10.1016/j.vaccine.2024.126273. Epub 2024 Sep 13. PMID 39276619

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 459 participants were enrolled, of which 454 were randomized and vaccinated in this study.
Groups:
- Cohort 1: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg): Participants received an intramuscular (IM) injection of Ad26/protein preF RSV vaccine composed of Ad26.RSV.preF at a dose level of 1*10^11 viral particles (vp) and RSV preF protein 150 microgram (mcg) on Day 1.
- Cohort 1: Ad26.RSV.preF (3.3*10^10 vp)+RSV preF Protein (150 mcg): Participants received an IM injection of Ad26/protein preF RSV vaccine composed of Ad26.RSV.preF at a dose level of 3.3*10^10 vp and RSV preF protein at a dose level of 150 mcg on Day 1.
- Cohort 1: Ad26.RSV.preF (1.1*10^10 vp)+RSV preF Protein (150 mcg): Participants received an IM injection of Ad26/protein preF RSV vaccine composed of Ad26.RSV.preF at a dose level of 1.1*10^10 vp and RSV preF protein at a dose level of 150 mcg on Day 1.
- Cohort 1: Ad26.RSV.preF (3.7*10^9 vp)+RSV preF Protein (150 mcg): Participants received an IM injection of Ad26/protein preF RSV vaccine composed of Ad26.RSV.preF at a dose level of 3.7*10^9 vp and RSV preF protein at a dose level of 150 mcg on Day 1.
- Cohort 1: Placebo; Cohort 2: Placebo; Cohort 3: Placebo: Participants received an IM injection of placebo matching to Ad26/protein preF RSV vaccine on Day 1.
- Cohort 2: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg); Cohort 3: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg): Participants received an IM injection of Ad26/protein preF RSV vaccine composed of Ad26.RSV.preF at a dose level of 1*10^11 vp and RSV preF protein at a dose level of 150 mcg on Day 1.
- Cohort 2: Ad26.RSV.preF (1.3*10^11 vp)+RSV preF Protein (150 mcg): Participants received an IM injection of Ad26/protein preF RSV vaccine composed of Ad26.RSV.preF at a dose level of 1.3*10^11 vp and RSV preF protein at a dose level of 150 mcg on Day 1.
- Cohort 3: Ad26.RSV.preF (1.6*10^11 vp)+RSV preF Protein (150 mcg): Participants received an IM injection of Ad26/protein preF RSV vaccine composed of Ad26.RSV.preF at a dose level of 1.6*10^11 vp and RSV preF protein at a dose level of 150 mcg on Day 1.
Period: Overall Study
Arm/Group | Cohort 1: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (3.3*10^10 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (1.1*10^10 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (3.7*10^9 vp)+RSV preF Protein (150 mcg) | Cohort 1: Placebo | Cohort 2: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 2: Ad26.RSV.preF (1.3*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 2: Placebo | Cohort 3: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 3: Ad26.RSV.preF (1.6*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 3: Placebo
Started | 51 | 51 | 51 | 48 | 25 | 49 | 49 | 26 | 27 | 51 | 26
Full Analysis Set (FAS) | 51 | 51 | 51 | 48 | 25 | 49 | 49 | 26 | 27 | 51 | 26
Per-protocol Immunogenicity (PPI) Set | 51 | 50 | 51 | 48 | 25 | 47 | 49 | 26 | 27 | 50 | 26
Completed | 50 | 48 | 50 | 45 | 24 | 47 | 48 | 26 | 27 | 48 | 25
Not Completed | 1 | 3 | 1 | 3 | 1 | 2 | 1 | 0 | 0 | 3 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (3.3*10^10 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (1.1*10^10 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (3.7*10^9 vp)+RSV preF Protein (150 mcg) | Cohort 1: Placebo | Cohort 2: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 2: Ad26.RSV.preF (1.3*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 2: Placebo | Cohort 3: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 3: Ad26.RSV.preF (1.6*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 3: Placebo | Total
Number analyzed (Participants) | 51 | 51 | 51 | 48 | 25 | 49 | 49 | 26 | 27 | 51 | 26 | 454
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (6.97) | 68.7 (7.08) | 69.4 (6.56) | 70.3 (6.82) | 70 (6.44) | 68.6 (6.69) | 68.6 (5.68) | 67.6 (5.34) | 67.9 (4.51) | 68.7 (5.41) | 66.5 (5.09) | 68.8 (6.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 30 | 25 | 14 | 17 | 29 | 16 | 16 | 28 | 10 | 247
  Male | 21 | 19 | 21 | 23 | 11 | 32 | 20 | 10 | 11 | 23 | 16 | 207
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 6 | 13 | 11 | 6 | 4 | 3 | 1 | 1 | 3 | 0 | 62
  Not Hispanic or Latino | 37 | 44 | 38 | 37 | 18 | 45 | 46 | 25 | 26 | 48 | 26 | 390
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Black or African American | 0 | 5 | 5 | 2 | 1 | 3 | 4 | 1 | 0 | 0 | 0 | 21
  White | 51 | 44 | 46 | 46 | 24 | 44 | 45 | 25 | 25 | 49 | 26 | 425
  More than one race | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 51 | 51 | 51 | 48 | 25 | 49 | 49 | 26 | 27 | 51 | 26 | 454

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Geometric Mean Antibody Titers to Respiratory Syncytial Virus (RSV) Prefusion Conformation-stabilized F (preF) Protein Using preF Enzyme-linked Immunosorbent Assay (ELISA) at 14 Days After Vaccination
Description: Geometric mean antibody titers (ELISA units per liter [EU/L]) to RSV preF protein using preF ELISA at 14 days after vaccination were reported.
Time Frame: 14 days after vaccination on Day 1 (Day 15)
Population: Per-protocol Immunogenicity (PPI) set included all participants who were randomized and received the study vaccine, and for whom immunogenicity data were available, excluding participants with major protocol deviations expecting to impact the immunogenicity outcomes. Here, 'N' (overall number of participants analyzed) signifies participants who were evaluated for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/L
Arm/Group | Cohort 1: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (3.3*10^10 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (1.1*10^10 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (3.7*10^9 vp)+RSV preF Protein (150 mcg) | Cohort 1: Placebo
Number analyzed (Participants) | 44 | 46 | 45 | 45 | 24
EU/L | 4907 [4030 to 5976] | 4681 [3696 to 5928] | 4038 [3042 to 5361] | 5238 [4070 to 6743] | 272 [212 to 350]

2. Primary Outcome: Cohorts 2 and 3: Number of Participants With Solicited Local Adverse Events (AEs) Until 7 Days After Vaccination on Day 1
Description: Number of participants with solicited local AEs until 7 days after vaccination on Day 1 were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs were pre-defined local (at the injection site) AEs for which participants were specifically questioned and which were noted by participants in their e-diary until 7 days after vaccination on Day 1 (day of vaccination and the subsequent 7 days). Solicited local AEs included: injection site pain/tenderness, erythema and swelling at the vaccination site.
Time Frame: Until 7 days after Vaccination on Day 1 (Day 8)
Population: Full Analysis Set (FAS) included all participants who were randomized and received the study vaccine, regardless of the occurrence of protocol deviations. Here, 'N' (overall number of participants analyzed) signifies participants who were evaluated for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 2: Ad26.RSV.preF (1.3*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 2: Placebo | Cohort 3: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 3: Ad26.RSV.preF (1.6*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 3: Placebo
Number analyzed (Participants) | 49 | 49 | 26 | 27 | 50 | 26
Participants | 37 | 42 | 3 | 23 | 37 | 2

3. Primary Outcome: Cohorts 2 and 3: Number of Participants With Solicited Systemic Adverse Events (AEs) Until 7 Days After Vaccination on Day 1
Description: Number of participants with solicited systemic AEs until 7 days after vaccination on Day 1 were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Participants were instructed on how to note signs and symptoms in their diary on a daily basis until 7 days post-vaccination (Day of vaccination and the subsequent 7 days) for solicited systemic AEs. Solicited systemic AEs included fatigue, headache, myalgia, nausea and fever (body temperature greater than or equal to [>=] 38 degree celsius).
Time Frame: Until 7 days after Vaccination on Day 1 (Day 8)
Population: FAS included all participants who were randomized and received the study vaccine, regardless of the occurrence of protocol deviations. Here, 'N' (overall number of participants analyzed) signifies participants who were evaluated for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 2: Ad26.RSV.preF (1.3*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 2: Placebo | Cohort 3: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 3: Ad26.RSV.preF (1.6*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 3: Placebo
Number analyzed (Participants) | 49 | 49 | 26 | 27 | 50 | 26
Participants | 39 | 43 | 8 | 19 | 41 | 7

4. Primary Outcome: Cohorts 2 and 3: Number of Participants With Unsolicited AEs Until 28 Days After Vaccination on Day 1
Description: Unsolicited AEs were all AEs for which the participants were not specifically questioned in the participant diary. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs included chills, injection site erythema, injection site pruritus Et cetera (etc).
Time Frame: Until 28 days after Vaccination on Day 1 (Day 29)
Population: FAS included all participants who were randomized and received the study vaccine, regardless of the occurrence of protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 2: Ad26.RSV.preF (1.3*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 2: Placebo | Cohort 3: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 3: Ad26.RSV.preF (1.6*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 3: Placebo
Number analyzed (Participants) | 49 | 49 | 26 | 27 | 51 | 26
Participants | 13 | 8 | 7 | 3 | 8 | 2

5. Secondary Outcome: Cohort 1: Geometric Mean Antibody Titers to RSV preF Protein Using preF ELISA at 3 and 6 Months After Vaccination on Day 1
Description: Geometric mean antibody titers (EU/L) to RSV preF protein using preF ELISA at 3 and 6 months after vaccination on Day 1 were reported.
Time Frame: At 3 and 6 months after vaccination on Day 1
Population: PPI set included all participants who were randomized and received the study vaccine, and for whom immunogenicity data were available, excluding participants with major protocol deviations expecting to impact the immunogenicity outcomes. Here, 'n' (number analyzed) signifies participants who were evaluable at specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/L
Arm/Group | Cohort 1: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (3.3*10^10 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (1.1*10^10 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (3.7*10^9 vp)+RSV preF Protein (150 mcg) | Cohort 1: Placebo
Number analyzed (Participants) | 51 | 50 | 51 | 48 | 25
EU/L
  3 months after vaccination on Day 1: number analyzed (Participants) | 51 | 48 | 51 | 45 | 24
  3 months after vaccination on Day 1 | 2550 [2134 to 3047] | 2790 [2251 to 3459] | 1940 [1565 to 2405] | 2997 [2335 to 3846] | 315 [251 to 394]
  6 months after vaccination on Day 1: number analyzed (Participants) | 48 | 45 | 46 | 42 | 23
  6 months after vaccination on Day 1 | 1568 [1351 to 1819] | 1424 [1126 to 1800] | 1247 [1053 to 1478] | 1834 [1478 to 2277] | 326 [256 to 414]

6. Secondary Outcome: Cohort 1: Respiratory Syncytial Virus (RSV) A2 Strain Neutralizing Antibody Titers at 14 Days and 3 and 6 Months After Vaccination on Day 1
Description: RSV A2 strain neutralizing antibody titers at 14 days and 3 and 6 months after vaccination on Day 1 were reported. RSV A2 strain neutralizing antibody titers of the vaccine-induced immune response was assessed through virus neutralization assay. Data were expressed as 50% inhibitory concentration (IC50) units.
Time Frame: At 14 days and 3 and 6 months after vaccination on Day 1
Population: PPI set included all participants who were randomized and received the study vaccine, and for whom immunogenicity data were available, excluding participants with major protocol deviations expecting to impact the immunogenicity outcomes. Here 'n' (number analyzed) signifies participants who were evaluable at specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 1: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (3.3*10^10 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (1.1*10^10 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (3.7*10^9 vp)+RSV preF Protein (150 mcg) | Cohort 1: Placebo
Number analyzed (Participants) | 51 | 50 | 51 | 48 | 25
Titer
  14 days after vaccination on Day 1: number analyzed (Participants) | 44 | 46 | 45 | 48 | 25
  14 days after vaccination on Day 1 | 6314 [4800 to 8307] | 5140 [3909 to 6758] | 4725 [3407 to 6554] | 6194 [4641 to 8265] | 294 [239 to 363]
  3 months after vaccination on Day 1: number analyzed (Participants) | 51 | 48 | 51 | 45 | 24
  3 months after vaccination on Day 1 | 3760 [2957 to 4780] | 3799 [2995 to 4820] | 2777 [2169 to 3556] | 4413 [3409 to 5713] | 357 [282 to 452]
  6 months after vaccination on Day 1: number analyzed (Participants) | 48 | 45 | 46 | 42 | 23
  6 months after vaccination on Day 1 | 1760 [1372 to 2260] | 1883 [1456 to 2435] | 1473 [1188 to 1827] | 2523 [1901 to 3348] | 301 [241 to 377]

7. Secondary Outcome: Cohort 1: T-cell Interferon (IFN) Gamma Responses to Respiratory Syncytial Virus (RSV) F Protein Peptides
Description: T-cell IFN gamma responses to RSV F protein specific peptides at 14 days and 3 and 6 months after vaccination as measured by enzyme-linked immunospot (ELISpot) assay were reported. RSV F specific T-cell IFN gamma ELISpot responses were measured as counts of spot forming cells per million peripheral blood mononuclear cells (SFC/10^6 PBMCs).
Time Frame: At 14 days and 3 and 6 months after vaccination on Day 1
Population: as for outcome 6
Measure: Median (Full Range); unit: SFC/10^6 PBMCs
Arm/Group | Cohort 1: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (3.3*10^10 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (1.1*10^10 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (3.7*10^9 vp)+RSV preF Protein (150 mcg) | Cohort 1: Placebo
Number analyzed (Participants) | 51 | 50 | 51 | 48 | 25
SFC/10^6 PBMCs
  14 days after vaccination on Day 1: number analyzed (Participants) | 37 | 42 | 36 | 36 | 19
  14 days after vaccination on Day 1 | 547 [NA to 1426] — Lower limit of full range could not be calculated as it was below the lower limit of quantification (LLOQ) (68) | 458 [NA to 1721] — Lower limit of full range could not be calculated as it was below the LLOQ (68) | 397 [79 to 1570] | 404 [87 to 1579] | NA [NA to 387] — Median lower limit of full range could not be calculated as it was below the LLOQ (68)
  3 months after vaccination on Day 1: number analyzed (Participants) | 46 | 46 | 47 | 38 | 22
  3 months after vaccination on Day 1 | 180 [NA to 1462] — Lower limit of full range could not be calculated as it was below the LLOQ (68). | 241 [NA to 906] — Lower limit of full range could not be calculated as it was below the LLOQ (68). | 168 [NA to 649] — Lower limit of full range could not be calculated as it was below the LLOQ (68). | 184 [NA to 737] — Lower limit of full range could not be calculated as it was below the LLOQ (68). | NA [NA to 359] — Median and lower limit of full range could not be calculated as it was below the LLOQ (68).
  6 months after vaccination on Day 1: number analyzed (Participants) | 45 | 44 | 45 | 42 | 23
  6 months after vaccination on Day 1 | 129 [NA to 1631] — Lower limit of full range could not be calculated as it was below the LLOQ (68). | 189 [NA to 991] — Lower limit of full range could not be calculated as it was below the LLOQ (68). | 146 [NA to 636] — Lower limit of full range could not be calculated as it was below the LLOQ (68). | 127 [NA to 439] — Lower limit of full range could not be calculated as it was below the LLOQ (68). | NA [NA to 266] — Median and lower limit of full range could not be calculated as it was below the LLOQ (68).

8. Secondary Outcome: Cohort 1: Number of Participants With Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was any untoward medical occurrence that at any dose resulted in death, was life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a suspected transmission of any infectious agent via a medicinal product.
Time Frame: Baseline (Day1) up to 6 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (3.3*10^10 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (1.1*10^10 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (3.7*10^9 vp)+RSV preF Protein (150 mcg) | Cohort 1: Placebo
Number analyzed (Participants) | 51 | 51 | 51 | 48 | 25
Participants | 3 | 0 | 0 | 1 | 0

9. Secondary Outcome: Cohort 1: Number of Participants With Solicited Local Adverse Events (AEs) Until 7 Days After Vaccination on Day 1
Description: as for outcome 2
Time Frame: Until 7 days after vaccination on Day 1 (Day 8)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (3.3*10^10 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (1.1*10^10 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (3.7*10^9 vp)+RSV preF Protein (150 mcg) | Cohort 1: Placebo
Number analyzed (Participants) | 51 | 50 | 51 | 47 | 25
Participants | 33 | 24 | 15 | 18 | 0

10. Secondary Outcome: Cohort 1: Number of Participants With Solicited Systemic Adverse Events (AEs) Until 7 Days After Vaccination on Day 1
Description: Number of participants with solicited systemic AEs until 7 days after vaccination on Day 1 were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Participants were instructed on how to note signs and symptoms in their diary on a daily basis until 7 days post-vaccination (Day of vaccination and the subsequent 7 days) for solicited systemic AEs. Solicited systemic AEs included fatigue, headache, myalgia, nausea and fever (body temperature >=38 degree celsius).
Time Frame: Until 7 days after vaccination on Day 1 (Day 8)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (3.3*10^10 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (1.1*10^10 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (3.7*10^9 vp)+RSV preF Protein (150 mcg) | Cohort 1: Placebo
Number analyzed (Participants) | 51 | 50 | 51 | 47 | 25
Participants | 35 | 25 | 13 | 15 | 6

11. Secondary Outcome: Cohort 1: Number of Participants With Unsolicited AEs Until 28 Days After Vaccination on Day 1
Description: Unsolicited AEs were all AEs for which the participants were not specifically questioned in the participant diary. Unsolicited AEs included chills, injection site erythema, injection site pruritus Et cetera (etc).
Time Frame: Until 28 days after vaccination on Day 1 (Day 29)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (3.3*10^10 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (1.1*10^10 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (3.7*10^9 vp)+RSV preF Protein (150 mcg) | Cohort 1: Placebo
Number analyzed (Participants) | 51 | 51 | 51 | 48 | 25
Participants | 11 | 9 | 6 | 5 | 1

12. Secondary Outcome: Cohort 2 and 3: Geometric Mean Antibody Titers to RSV preF Protein Using preF ELISA at 14 Days and 3 and 6 Months After Vaccination on Day 1
Description: Geometric mean antibody titers (EU/L) to RSV preF protein using preF ELISA at 14 days and 3 and 6 months after vaccination on Day 1 were reported.
Time Frame: At 14 days and 3 and 6 months after vaccination on Day 1
Population: PPI set was analyzed. Here, 'N' (overall number of participants analyzed) signifies participants who were evaluated for this outcome measure. Here 'n' (number analyzed) signifies participants who were evaluable at specified time points. Due to change in planned analysis, data at 6-month was not collected and analyzed because of discontinuation of the development of the vaccine and hence, there was no scientific value to analyze the responses at Month 6.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/L
Arm/Group | Cohort 2: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 2: Ad26.RSV.preF (1.3*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 2: Placebo | Cohort 3: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 3: Ad26.RSV.preF (1.6*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 3: Placebo
Number analyzed (Participants) | 45 | 49 | 26 | 26 | 47 | 26
EU/L
  14 days after vaccination on Day 1 | 3769 [3006 to 4726] | 3893 [3243 to 4674] | 259 [201 to 333] | 4278 [3336 to 5486] | 3856 [3177 to 4682] | 298 [236 to 376]
  3 months after vaccination on Day 1: number analyzed (Participants) | 44 | 47 | 26 | 26 | 47 | 26
  3 months after vaccination on Day 1 | 1982 [1627 to 2415] | 1665 [1162 to 2385] | 300 [244 to 369] | 2696 [1991 to 3651] | 1864 [1304 to 2664] | 339 [256 to 450]

13. Secondary Outcome: Cohort 2 and 3: Respiratory Syncytial Virus (RSV) A2 Strain Neutralizing Antibody Titers at 14 Days and 3 and 6 Months After Vaccination on Day 1
Description: RSV A2 neutralizing antibody titers at 14 days and 3 and 6 months after vaccination on Day 1 were reported. RSV A2 strain neutralizing antibody titers of the vaccine-induced immune response was assessed through virus neutralization assay. Data were expressed as 50% IC50 units.
Time Frame: At 14 days and 3 and 6 months after vaccination on Day 1
Population: PPI set included all participants who were randomized and received the study vaccine, and for whom immunogenicity data were available, excluding participants with major protocol deviations expecting to impact the immunogenicity outcomes. Here, 'N' (overall number of participants analyzed) signifies participants who were evaluated for this outcome measure. Here 'n' (number analyzed) signifies participants who were evaluable at specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 2: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 2: Ad26.RSV.preF (1.3*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 2: Placebo | Cohort 3: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 3: Ad26.RSV.preF (1.6*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 3: Placebo
Number analyzed (Participants) | 45 | 49 | 26 | 26 | 47 | 26
Titer
  14 days after vaccination on Day 1 | 4102 [3064 to 5491] | 3552 [2635 to 4789] | 336 [262 to 432] | 4085 [3092 to 5398] | 3707 [2841 to 4839] | 342 [261 to 448]
  3 months after vaccination on Day 1: number analyzed (Participants) | 44 | 47 | 26 | 25 | 47 | 26
  3 months after vaccination on Day 1 | 3144 [2537 to 3895] | 2556 [1828 to 3575] | 371 [282 to 488] | 3435 [2714 to 4348] | 2671 [1945 to 3669] | 490 [344 to 698]
  6 months after vaccination on Day 1: number analyzed (Participants) | 40 | 44 | 24 | 25 | 47 | 25
  6 months after vaccination on Day 1 | 1983 [1352 to 2909] | 1890 [1460 to 2447] | 356 [270 to 470] | 2168 [1682 to 2794] | 1856 [1509 to 2283] | 356 [274 to 464]

14. Secondary Outcome: Cohort 2 and 3: T-cell Interferon (IFN) Gamma Responses to Respiratory Syncytial Virus (RSV) F Protein Peptides at 14 Days and 3 and 6 Months After Vaccination on Day 1
Description: T-cell IFN gamma responses to RSV F protein specific peptides at 14 days and 3 and 6 months after vaccination as measured by ELISpot assay were reported. RSV F specific T-cell IFN gamma ELISpot responses were measured as counts of spot forming cells per million peripheral blood mononuclear cells (SFC/10^6 PBMCs).
Time Frame: At 14 days and 3 and 6 months after vaccination on Day 1
Population: PPI set was analyzed. Here, 'N' (overall number of participants analyzed) signifies participants evaluated for this outcome measure. Here 'n' (number analyzed) signifies number of participants evaluable at specified time points. Due to change in planned analysis, data at 6-month was not collected and analyzed because of discontinuation of the development of the vaccine and hence, there was no scientific value to analyze the responses at Month 6.
Measure: Median (Full Range); unit: SFC/10^6 PBMCs
Arm/Group | Cohort 2: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 2: Ad26.RSV.preF (1.3*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 2: Placebo | Cohort 3: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 3: Ad26.RSV.preF (1.6*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 3: Placebo
Number analyzed (Participants) | 40 | 42 | 22 | 25 | 45 | 24
SFC/10^6 PBMCs
  14 days after vaccination on Day 1: number analyzed (Participants) | 40 | 42 | 21 | 19 | 41 | 20
  14 days after vaccination on Day 1 | 361 [NA to 1686] — Lower limit of full range could not be calculated as it was below the LLOQ (68). | 435 [88 to 2088] | NA [NA to 942] — Median and lower limit of full range could not be calculated as it was below the LLOQ (68). | 236 [NA to 1764] — Lower limit of full range could not be calculated as it was below the LLOQ (68). | 204 [NA to 1888] — Lower limit of full range could not be calculated as it was below the LLOQ (68). | NA [NA to 216] — Median and lower limit of full range could not be calculated as it was below the LLOQ (68).
  3 months after vaccination on Day 1: number analyzed (Participants) | 37 | 40 | 22 | 25 | 45 | 24
  3 months after vaccination on Day 1 | 331 [NA to 1287] — Lower limit of full range could not be calculated as it was below the LLOQ (68). | 274 [NA to 1831] — Lower limit of full range could not be calculated as it was below the LLOQ (68). | NA [NA to 376] — Median and lower limit of full range could not be calculated as it was below the LLOQ (68). | 131 [NA to 851] — Lower limit of full range could not be calculated as it was below the LLOQ (68). | 172 [NA to 2737] — Lower limit of full range could not be calculated as it was below the LLOQ (68). | NA [NA to 212] — Median and lower limit of full range could not be calculated as it was below the LLOQ (68).

15. Secondary Outcome: Cohort 2 and 3: Number of Participants With Serious Adverse Events (SAEs)
Description: as for outcome 8
Time Frame: Baseline (Day1 ) up to 6 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 2: Ad26.RSV.preF (1.3*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 2: Placebo | Cohort 3: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 3: Ad26.RSV.preF (1.6*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 3: Placebo
Number analyzed (Participants) | 49 | 49 | 26 | 27 | 51 | 26
Participants | 1 | 1 | 1 | 0 | 2 | 1

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to 6 months
Description: FAS included all participants who were randomized and received the study vaccine, regardless of the occurrence of protocol deviations.
Arm/Group | Cohort 1: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (3.3*10^10 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (1.1*10^10 vp)+RSV preF Protein (150 mcg) | Cohort 1: Ad26.RSV.preF (3.7*10^9 vp)+RSV preF Protein (150 mcg) | Cohort 1: Placebo | Cohort 2: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 2: Ad26.RSV.preF (1.3*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 2: Placebo | Cohort 3: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 3: Ad26.RSV.preF (1.6*10^11 vp)+RSV preF Protein (150 mcg) | Cohort 3: Placebo
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51 | 0/51 | 0/48 | 0/25 | 0/49 | 0/49 | 0/26 | 0/27 | 1/51 | 0/26
Serious Adverse Events (participants affected / at risk) | 3/51 | 0/51 | 0/51 | 1/48 | 0/25 | 1/49 | 1/49 | 1/26 | 0/27 | 2/51 | 1/26
Other Adverse Events (participants affected / at risk) | 42/51 | 36/51 | 25/51 | 23/48 | 7/25 | 44/49 | 48/49 | 13/26 | 25/27 | 44/51 | 8/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) (N=51) | Cohort 1: Ad26.RSV.preF (3.3*10^10 vp)+RSV preF Protein (150 mcg) (N=51) | Cohort 1: Ad26.RSV.preF (1.1*10^10 vp)+RSV preF Protein (150 mcg) (N=51) | Cohort 1: Ad26.RSV.preF (3.7*10^9 vp)+RSV preF Protein (150 mcg) (N=48) | Cohort 1: Placebo (N=25) | Cohort 2: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) (N=49) | Cohort 2: Ad26.RSV.preF (1.3*10^11 vp)+RSV preF Protein (150 mcg) (N=49) | Cohort 2: Placebo (N=26) | Cohort 3: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) (N=27) | Cohort 3: Ad26.RSV.preF (1.6*10^11 vp)+RSV preF Protein (150 mcg) (N=51) | Cohort 3: Placebo (N=26)
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Covid-19 Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) (N=51) | Cohort 1: Ad26.RSV.preF (3.3*10^10 vp)+RSV preF Protein (150 mcg) (N=51) | Cohort 1: Ad26.RSV.preF (1.1*10^10 vp)+RSV preF Protein (150 mcg) (N=51) | Cohort 1: Ad26.RSV.preF (3.7*10^9 vp)+RSV preF Protein (150 mcg) (N=48) | Cohort 1: Placebo (N=25) | Cohort 2: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) (N=49) | Cohort 2: Ad26.RSV.preF (1.3*10^11 vp)+RSV preF Protein (150 mcg) (N=49) | Cohort 2: Placebo (N=26) | Cohort 3: Ad26.RSV.preF (1*10^11 vp)+RSV preF Protein (150 mcg) (N=27) | Cohort 3: Ad26.RSV.preF (1.6*10^11 vp)+RSV preF Protein (150 mcg) (N=51) | Cohort 3: Placebo (N=26)
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 6 | 2 | 0 | 2 | 5 | 13 | 2 | 6 | 10 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 3 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 2 | 0
Fatigue (General disorders) | 29 | 16 | 10 | 12 | 5 | 32 | 37 | 4 | 16 | 34 | 7
Influenza Like Illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection Site Haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection Site Pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0 | 0 | 6 | 11 | 1 | 4 | 12 | 0
Swelling (General disorders) | 2 | 6 | 2 | 3 | 0 | 7 | 7 | 0 | 2 | 9 | 0
Swelling Face (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tenderness (General disorders) | 32 | 23 | 12 | 17 | 0 | 34 | 40 | 2 | 23 | 37 | 2
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Pressure Systolic Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 21 | 12 | 4 | 5 | 1 | 25 | 29 | 1 | 17 | 23 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 18 | 12 | 6 | 2 | 3 | 25 | 25 | 2 | 15 | 27 | 3
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Taste Disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vith Nerve Paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Adjustment Disorder with Depressed Mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Respiratory Symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 6 | 4 | 2 | 1 | 0 | 7 | 7 | 1 | 2 | 9 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/02/NCT04453202/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/02/NCT04453202/SAP_001.pdf